CLINICAL TRIAL: NCT06454955
Title: Study of B7-H3 Mediated Tumor Immune Response Using a Whole-Body Kinetic Approach in Whole-Body PET
Brief Title: Study on B7-H3 Targeted Affibody Radioligand Probes for PET Imaging of Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023KT131
Record Dates: First submitted 2024-05-30; First posted 2024-06-12 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-01

CONDITIONS: B7H3; CD276 Affibody; PET/CT Imaing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Each patient must undergo dynamic PET/CT imaging with [68Ga]B7H3 Affibody-BCH. (Experimental)
  Interventions: Drug: [68Ga] B7H3 Affibody-BCH

INTERVENTIONS:
Drug: [68Ga] B7H3 Affibody-BCH — An affibody structure specifically targeting B7H3 was developed based on the B7H3 binding domain, and it was structurally optimized to yield a small molecular agent, B7H3 Affibody-BCH, suitable for nuclear medical diagnostic and therapeutic uses targeting B7H3. By labeling with the radioactive isotope ^68Ga, this agent can be used for PET/CT diagnosis of solid tumors.

SUMMARY:
Based on [68Ga]B7H3 Affibody-BCH, this study investigates its radioactive uptake and imaging capabilities in tumor patients, with the aim of establishing a correlation between radioactive uptake and B7-H3 receptor expression. Utilizing whole-body PET technology, the pharmacokinetic dynamics of [68Ga]B7H3 Affibody-BCH are examined to ascertain its pharmacological characteristics. Ultimately, this research establishes a framework for pharmacokinetic analysis using whole-body PET.

ELIGIBILITY:
Inclusion Criteria:

1. Age range 18-75 years, open to both male and female participants;
2. Participants must meet the following hematologic and hepatic/renal function criteria: Hematology: WBC ≥ 4.0 × 10^9/L or neutrophils ≥ 1.5 × 10^9/L, platelets ≥ 100 × 10^9/L, hemoglobin ≥ 90 g/L; Prothrombin time (PT) or Activated partial thromboplastin time (APTT) ≤ 1.5 times the upper limit of normal (ULN); Hepatic and renal functions: Total bilirubin (T-Bil) ≤ 1.5 times the upper threshold limit (ULT), ALT/AST ≤ 2.5 ULN or ≤ 5 ULT for subjects with liver metastasis, Alkaline phosphatase (ALP) ≤ 2.5 ULN (or ≤ 4.5 ULN in cases of bone or liver metastasis); Blood urea nitrogen (BUN) ≤ 1.5 × ULT, serum creatinine (SCr) ≤ 1.5 × ULT;
3. Normal cardiac function;
4. Expected survival of at least 12 weeks;
5. Good adherence to follow-up;
6. Presence of at least one measurable target lesion according to RECIST 1.1 criteria;
7. Women of childbearing age (15-49 years) must undergo a pregnancy test within seven days prior to the commencement of the study and test negative; sexually active male and female participants must agree to utilize effective contraception to prevent pregnancy during the study and for three months following the final examination;
8. Patients for whom a clinical physician recommends PET/CT scans for the diagnosis and staging of tumors;
9. Participants must fully understand and voluntarily agree to participate in the study, and must sign an informed consent form.

Exclusion Criteria:

1. Severe abnormalities in liver and renal function and blood counts;
2. Patients planning to conceive;
3. Pregnant or lactating women;
4. Individuals unable to lie flat for thirty minutes;
5. Individuals who refuse to participate in this clinical study;
6. Individuals suffering from claustrophobia or other psychiatric disorders;
7. Other situations deemed unsuitable for trial participation by the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
SUV | 1 hour and 2 hour after injection
  Standardized Uptake Values (SUV) of [68Ga] B7H3 Affibody-BCH at various time points within the imaging window for target lesions or suspected tumor lesions in subjects with malignant tumors.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangxi Meng, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Xia L, Wu Y, Ren Y, Wang Z, Zhou N, Zhou W, Zhou L, Jia L, He C, Meng X, Zhu H, Yang Z. A whole-body imaging technique for tumor-specific diagnostics and screening of B7H3-targeted therapies. J Clin Invest. 2025 Jan 23;135(6):e186388. doi: 10.1172/JCI186388. PMID 39847434